CLINICAL TRIAL: NCT02289430
Title: A Phase I Clinical Trial to Investigate the Pharmacokinetic Interactions and Safety Between Rosuvastatin and Ezetimibe in Healthy Male Volunteers
Brief Title: to Investigate the Pharmacokinetic Interactions and Safety Between Rosuvastatin and Ezetimibe in Healthy Male Volunteers
Acronym: NVP-1205
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NVP Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NVP-1205-02
Record Dates: First submitted 2014-11-09; First posted 2014-11-13 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
MeSH Terms: interventions — Ezetimibe; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Crestor+Ezetrol (Experimental): rosuvastatin+ezetimibe
  Interventions: Drug: Crestor+Ezetrol
- Ezetrol (Active Comparator): ezetimibe
  Interventions: Drug: Ezetrol
- Crestor (Active Comparator): rosuvastatin
  Interventions: Drug: Crestor

INTERVENTIONS:
Drug: Crestor+Ezetrol — rosuvastatin+ezetimibe
  Other Names: rosuvatatin+ezetimibe
  Arms: Crestor+Ezetrol
Drug: Ezetrol — ezetimibe
  Other Names: ezetimibe
  Arms: Ezetrol
Drug: Crestor — rosuvastatin
  Other Names: rosuvastatin
  Arms: Crestor

SUMMARY:
The purpose of this study is to compare the drug interaction of pharmacokinetics of rosuvastatin and ezetimibe.

DETAILED DESCRIPTION:
drug interaction : rosuvastatin, ezetimibe

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects age between 19 and 45 singed informed consent

Exclusion Criteria:

* Hypotension or hypertension has a history of allergy reaction of this drug or other drugs

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2014-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Area Under Curve | 0-24h

CONTACTS AND LOCATIONS:
Overall Officials: Shin D Seong, M.D., Principal Investigator — Gachon University Gil Medical Center

IPD SHARING:
Plan to Share IPD: No